CLINICAL TRIAL: NCT06822244
Title: The Effect of Pranayama Exercise on Vital Signs, Anxiety, Fear of Death, and Sleep Quality After Acute Myocardial Infarction
Brief Title: The Effect of Pranayama Exercise
Acronym: Pranayama
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Berna Dincer, Nursing Associate Professor, Istanbul Medeniyet University
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IstanbulMU; 00144 (Other Grant/Funding Number: medeniyet university)
Record Dates: First submitted 2025-01-30; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pranayama; Exercise; Anxiety; Death; Sleep
Keywords: pranayama; Exercise; Anxiety; Death; Sleep
MeSH Terms: conditions — Motor Activity; Anxiety Disorders; Death

STUDY DESIGN:
Intervention Model Description: Assuming a power of 80% and an α risk of. 05, a sample size of 75 was determined to be appropriate. Considering the possibility of missing data, the study initially included 80 participants in both the experimental and control groups. A computer-based random number generator was used for group assignment, and allocation concealment was ensured by using sealed envelopes containing random numbers opened by a separate researcher. The study was completed with 40 participants in the experimental group and 40 in the control group, due to some participants withdrawing.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pranayama exercise (Experimental): Do Pranayama Exercise
  Interventions: Behavioral: Pranayama exercise
- Control (Active Comparator): do Nothing
  Interventions: Behavioral: normal breathing

INTERVENTIONS:
Behavioral: Pranayama exercise — The people in the pranayama experimental group were first informed about the practice (At the deepest point of the breath, the left nostril is closed with the index finger of the right hand and exhaled through the right nostril. When it reaches the deepest point, close the nostril with the thumb and exhale through the left nostril. At least 3 more rounds are continued in this way.
  one Pranayama session (approximately 30 minutes). The people in the experimental group were taught pranayama exercises during the application and were given a brochure with written instructions on home application and were info
  Arms: Pranayama exercise
Behavioral: normal breathing — normal breathing 20 breath per min
  Arms: Control

SUMMARY:
Objective: This randomized controlled experimental study aimed to investigate the effects of pranayama exercises on vital signs, anxiety, fear of death, and sleep quality in patients who have experienced an acute myocardial infarction.

Materials and Methods: The study sample consisted of 80 patients diagnosed with acute myocardial infarction who were hospitalized in the Coronary Intensive Care Unit of Istanbul University Cerrahpaşa Medical Faculty Hospital The patients were randomly assigned to either the experimental (n=40) or control group (n=40) using a computer-based randomization method. Data collection tools included the Personal Information Form, Beck Anxiety Inventory, Death Anxiety Scale, and Pittsburgh Sleep Quality Index.

DETAILED DESCRIPTION:
Objective: This randomized controlled experimental study aimed to investigate the effects of pranayama exercises on vital signs, anxiety, fear of death, and sleep quality in patients who have experienced an acute myocardial infarction.

Materials and Methods: The study sample consisted of 80 patients diagnosed with acute myocardial infarction who were hospitalized in the Coronary Intensive Care Unit of Istanbul University Cerrahpaşa Medical Faculty Hospital between June and November 2024. The patients were randomly assigned to either the experimental (n=40) or control group (n=40) using a computer-based randomization method. Data collection tools included the Personal Information Form, Beck Anxiety Inventory, Death Anxiety Scale, and Pittsburgh Sleep Quality Index.

ELIGIBILITY:
Inclusion Criteria:

Voluntary participation in the study

Age ≥18 years

Diagnosed with AMI

Cognitive ability to perform pranayama exercises

Ability to comprehend and respond to survey questions

No communication impairments

Exclusion Criteria:

* having respiratory diseases
* low saturation <95

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory | up to 4 weeks
  It is a Likert-type scale consisting of 21 items and scored between 0-3. According to scale scoring; 8 points: No anxiety, 8-15 points: Mild anxiety, 16-25 points: Moderate anxiety, 26-63 points: Determined as severe anxiety decrease the15 points

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No